CLINICAL TRIAL: NCT02674386
Title: A PHASE 3, MULTICENTER, LONG-TERM OBSERVATIONAL STUDY OF SUBJECTS FROM TANEZUMAB STUDIES WHO UNDERGO A TOTAL KNEE, HIP OR SHOULDER REPLACEMENT
Brief Title: Long-term Observational Study of Subjects From Tanezumab Studies Who Undergo a Total Knee, Hip or Shoulder Replacement
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: A4091064; 2013-002549-12 (EudraCT Number); TJR FOLLOW-UP (Other: Alias Study Number)
Record Dates: First submitted 2015-11-11; First posted 2016-02-04 (Estimated); Results first posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Inosine Monophosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cohort 1 (Other): long-term observational study of subjects from tanezumab parent study
  Interventions: Drug: Investigational Medical Product (IMP) administered in parent study

INTERVENTIONS:
Drug: Investigational Medical Product (IMP) administered in parent study — IMP as administered in parent study. IMP would have been either placebo, tanezumab, celecoxib, naproxen or diclofenac administered in parent study.

SUMMARY:
A4091064 is a multicenter, long-term observational study of subjects from tanezumab interventional studies (regardless of treatment group) who undergo a total knee, hip or shoulder replacement during participation in the study. The study is designed with a total duration of subject follow-up of 24 weeks after the total joint replacement surgery. There will be two methods of data collection utilized in this study: interview by site staff via the telephone and interactive web-response system (or paper if the subject has no access to the internet).

DETAILED DESCRIPTION:
A4091064 is a long-term observational follow up study of subjects from tanezumab interventional studies A4091056, A4091057 or A4091058.

ELIGIBILITY:
Inclusion Criteria:

* Personally signed and dated informed consent document.
* Randomized and treated with subcutaneous investigational product in a tanezumab study and has completed the study or been withdrawn from the study.
* Actual or planned total knee, hip or shoulder replacement surgery during the tanezumab study.
* Willing and able to comply with scheduled visits and other study procedures.

Exclusion Criteria:

- None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2016-08-23 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (79):
- United States (51):
  - Central Alabama Research, Birmingham, Alabama
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Alabama Orthopaedic Surgeons, Birmingham, Alabama
  - Cahaba Research Inc., Birmingham, Alabama
  - Noble Clinical Research, Tucson, Arizona
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - Advanced Research Center, Inc., Anaheim, California
  - Hope Clinical Research, Canoga Park, California
  - Marvel Clinical Research, LLC, Huntington Beach, California
  - Advances in Medicine, Palm Desert, California
  - Clinical Trials Research, Sacramento, California
  - California Research Foundation, San Diego, California
  - CITrials, Santa Ana, California
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - JEM Research Institute, Atlantis, Florida
  - Orthopedic Research Institute, Boynton Beach, Florida
  - Orthopaedic Associates of West Florida, Clearwater, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Clintex Research Group, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - American Family Medical, Ocala, Florida
  - Sunshine Research Center, Opa-locka, Florida
  - Gulfcoast Research Institute, LLC, Sarasota, Florida
  - Kennedy White Orthopaedic Center, Sarasota, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Masters of Clinical Research, Inc., Augusta, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - North Georgia Internal Medicine, Woodstock, Georgia
  - Injury Care Research, Boise, Idaho
  - Chicago Clinical Research Institute, Inc., Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Professional Research Network of Kansas, LLC, Wichita, Kansas
  - Best Clinical Trials, LLC, New Orleans, Louisiana
  - George Stanley Walker, MD, New Orleans, Louisiana
  - Great Lakes Research Group, Incorporated, Bay City, Michigan
  - Orthopaedic Associates of Michigan, PC, Grand Rapids, Michigan
  - Physician Research Collaboration, LLC, Lincoln, Nebraska
  - Drug Trials America, Hartsdale, New York
  - Remington-Davis, Incorporated, Columbus, Ohio
  - Optimed Research LTD, Columbus, Ohio
  - AC Clinical Research, Tiffin, Ohio
  - Founders Research Corporation, Philadelphia, Pennsylvania
  - Abigail R. Neiman, MD, PA, Houston, Texas
  - Advances In Health, Houston, Texas
  - Mercury Clinical Research, Inc., Houston, Texas
  - BI Research Center, Houston, Texas
  - ClinRx Research, Richardson, Texas
  - DCT - Stone Oak, LLC dba Discovery Clinical Trials, San Antonio, Texas
  - Mercury Clinical Research, Webster, Texas
  - Spectrum Medical, Inc., Danville, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
- CMAX Clinical Research Pty Ltd, Adelaide, South Australia, Australia
- Canada (4):
  - Dawson Road Medical Centre, Guelph, Ontario
  - Rebecca Medical Associates, Oakville, Ontario
  - Recherche Clinique Sigma inc, Québec, Quebec
  - Centre de recherche Saint-Louis, Québec, Quebec
- Rheumazentrum Prof. Dr. med Gunther Neeck, Bad Doberan, Germany
- Tolna Megyei Balassa Janos Korhaz, Ortopediai Osztaly, Szekszárd, Hungary
- Azienda Ospedaliero-Universitaria E Policlinico Umberto I, Rome, Italy
- Japan (5):
  - Omuro Orthopedic Clinic, Himeji, Hyōgo
  - Nakajo Orthopedic Clinic, Sendai, Miyagi
  - Marunouchi Hospital, Matsumoto, Nagano
  - National Hospital Organization Osaka Minami Medical Center, Kawachi-Nagano, Osaka
  - Osaka University Hospital, Suita, Osaka
- Saules seimos medicinos centras, Kaunas, Lithuania
- New Zealand (4):
  - South Pacific Clinical Trials, Auckland
  - Star Unit, North Shore Hospital, Waitemata District Health Board, Auckland
  - Southern Clinical Trials- Waitemata Ltd, Auckland
  - Clinical Horizons NZ Ltd, Tauranga
- Hospital Conde de Bertiandos, Ponte de Lima, Viana do Castelo District, Portugal
- Medical Technologies Ltd., Saint Petersburg, Russia
- Institute of Rheumatology, Belgrade, Serbia
- Slovakia (2):
  - Kompan, s.r.o., Dolný Kubín
  - Slovak Research Center Team Member, MUDr. Viliam Cibik, PhD, s.r.o., Pruské
- Spain (2):
  - Instituto de Ciencias Medicas, Alicante
  - Hospital del Mar, Barcelona
- Sweden (3):
  - Ladulaas Kliniska Studier, Boras, Sweden
  - ProbarE I Lund AB, Lund
  - ProbarE i Stockholm AB, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Mont MA, Carrino JA, Nemeth MA, Burr A, Yamabe T, Viktrup L, Brown MT, West CR, Verburg KM. Postoperative Outcome of Patients Who Underwent Total Joint Replacement During the Tanezumab Phase 3 Osteoarthritis Development Program: A 24-Week Observational Study. Surg Technol Int. 2021 May 20;38:467-477. doi: 10.52198/21.STI.38.OS1439. PMID 34043229
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A4091064

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study included participants from studies A4091056 (NCT02697773), A4091057 (NCT02709486) and A4091058 (NCT02528188) who had undergone a total joint replacement (TJR) surgery of knee, hip, or shoulder. During this study, if participant underwent an additional TJR surgery, then data for that additional TJR surgery was also assessed.
Pre-assignment Details: Pre-specified intent of this study was to compare results regardless of treatment group/doses in parent studies and also to report data for overall (combined participants from all parent studies).
Groups:
- Placebo: Participants who received placebo matched to tanezumab in studies A4091056 (NCT02697773) and A4091057 (NCT02709486) and who had undergone a TJR surgery, were followed up for a maximum duration of 24 weeks in this study. Baseline for this study was the last visit in study A4091056, A4091057 or A4091058 (NCT02528188) or when the site notified of a planned TJR surgery.
- Tanezumab Combined: Participants who received tanezumab subcutaneous (SC) injection of 2.5 milligram (mg) or 2.5 mg/5 mg or 5 mg in studies A4091056, A4091057 or A4091058 and who had undergone a TJR surgery, were followed up for a maximum duration of 24 weeks in this study. Baseline for this study was the last visit in study A4091056, A4091057 or A4091058 or when the site notified of a planned TJR surgery.
- NSAID: Participants who received non-steroidal anti-inflammatory drug (NSAID) tablets (naproxen 500 mg, celecoxib 100 mg, or diclofenac extended release 75 mg) in study A4091058 and who had undergone a TJR surgery, were followed up for a maximum duration of 24 weeks in this study. Baseline for this study was the last visit in study A4091056, A4091057 or A4091058 or when the site notified of a planned TJR surgery.
Period: Overall Study
Arm/Group | Placebo | Tanezumab Combined | NSAID
Started | 20 | 117 | 17
Safety Analysis Set | 20 | 113 | 17
Completed | 20 | 107 | 16
Not Completed | 0 | 10 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 4 | 0
Not completed — Other | 0 | 1 | 0
Not completed — Enrolled but not evaluated | 0 | 4 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set: all enrolled participants of this study who had received at least one dose of SC study medication during studies A4091056, A4091057 or A4091058, and who had a qualifying i.e. total (not partial) joint replacement surgery.
Groups:
- Tanezumab Combined: Participants who received tanezumab SC injection of 2.5 mg or 2.5 mg/5 mg or 5 mg in studies A4091056, A4091057 or A4091058 and who had undergone a TJR surgery, were followed up for a maximum duration of 24 weeks in this study. Baseline for this study was the last visit in study A4091056, A4091057 or A4091058 or when the site notified of a planned TJR surgery.
- NSAID: Participants who received NSAID tablets (naproxen 500 mg, celecoxib 100 mg, or diclofenac extended release 75 mg) in study A4091058 and who had undergone a TJR surgery, were followed up for a maximum duration of 24 weeks in this study. Baseline for this study was the last visit in study A4091056, A4091057 or A4091058 or when the site notified of a planned TJR surgery.
- Total: Total of all reporting groups
Arm/Group | Placebo | Tanezumab Combined | NSAID | Total
Number analyzed (Participants) | 20 | 113 | 17 | 150
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.26 (8.77) | 64.57 (8.18) | 62.94 (9.13) | 64.47 (8.33)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 6 | 50 | 4 | 60
  Female | 13 | 62 | 13 | 88
  Unspecified | 1 | 1 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 3 | 7
  Not Hispanic or Latino | 18 | 109 | 14 | 141
  Unknown or Not Reported | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 6 | 0 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 6 | 3 | 9
  White | 17 | 100 | 14 | 131
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Surgeon's Assessment of Procedural Difficulty
Description: Following the TJR surgery on Day 1, the orthopedic surgeon was asked to answer the following question: "taking into consideration the participant's medical history and physical condition prior to surgery would you classify the operative procedure as Uneventful, Minor complications or Major complications." Participants were reported based on these categories for knee, hip and shoulder joint. Participants may have been counted more than once if they had TJR surgery in more than one joint.
Time Frame: Day 1
Population: Safety analysis set analyzed. Here, 'Overall number of participants analyzed (N)' = only those participants who had data available for this outcome measure (OM). 'Number analyzed (n)' = participants evaluable for this OM at specified categories.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: All participants who received placebo matched to tanezumab in studies A4091056 and A4091057; received tanezumab SC injection of 2.5 mg or 2.5 mg/5 mg or 5 mg in studies A4091056, A4091057 or A4091058 and who received NSAID tablets (naproxen 500 mg, celecoxib 100 mg, or diclofenac extended release 75 mg) in study A4091058 and who had undergone a TJR surgery.
Arm/Group | Placebo | Tanezumab Combined | NSAID | All Participants
Number analyzed (Participants) | 17 | 92 | 13 | 122
Participants
  Knee: number analyzed (Participants) | 9 | 51 | 8 | 68
  Knee: Uneventful | 9 | 49 | 8 | 66
  Knee: Minor Complications | 0 | 2 | 0 | 2
  Knee: Major Complications | 0 | 0 | 0 | 0
  Hip: number analyzed (Participants) | 8 | 41 | 4 | 53
  Hip: Uneventful | 8 | 37 | 4 | 49
  Hip: Minor Complications | 0 | 4 | 0 | 4
  Hip: Major Complications | 0 | 0 | 0 | 0
  Shoulder: number analyzed (Participants) | 0 | 0 | 1 | 1
  Shoulder: Uneventful | 0 | 0 | 1 | 1
  Shoulder: Minor Complications | 0 | 0 | 0 | 0
  Shoulder: Major Complications | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Overall Satisfaction With Surgery as Assessed by the Self-Administered Patient Satisfaction (SAPS) Scale at Week 24
Description: SAPS contained four questions; How satisfied are you with the 1) results of your surgery 2) results of surgery for improving pain 3) results of surgery for improving ability to do home or yard work, and 4) results of surgery for improving your ability to do recreational activities. Items scored on a 4-point Likert scale with response of 'very satisfied' (100 points), 'somewhat satisfied' (75 points), 'somewhat dissatisfied' (50 points), and 'very dissatisfied' (25 points). The scale score calculated as mean of the scores of individual items, ranging from 25 to 100, with higher scores indicating greater satisfaction. Here, number of participants are summarized as, satisfied (very satisfied and somewhat satisfied categories combined) and dissatisfied (somewhat dissatisfied and very dissatisfied categories combined). Participants may have been counted more than once if they had TJR surgery in more than one joint.
Time Frame: Week 24
Population: Safety analysis set: enrolled participants who had received at least one dose of SC study medication during studies A4091056, A4091057 or A4091058, and who had a qualifying TJR surgery. Here, 'N' signifies only those participants who had data available for this OM. 'n' = participants evaluable for this OM at specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab Combined | NSAID | All Participants
Number analyzed (Participants) | 19 | 99 | 13 | 131
Participants
  Knee: Satisfaction with result of surgery: number analyzed (Participants) | 9 | 58 | 6 | 73
  Knee: Satisfaction with result of surgery: Satisfied | 9 | 53 | 5 | 67
  Knee: Satisfaction with result of surgery: Dissatisfied | 0 | 5 | 1 | 6
  Knee: Results of surgery for relieving pain: number analyzed (Participants) | 9 | 58 | 6 | 73
  Knee: Results of surgery for relieving pain: Satisfied | 9 | 52 | 5 | 66
  Knee: Results of surgery for relieving pain: Dissatisfied | 0 | 6 | 1 | 7
  Knee: Improving ability for home or yard work: number analyzed (Participants) | 9 | 58 | 6 | 73
  Knee: Improving ability for home or yard work: Satisfied | 9 | 48 | 5 | 62
  Knee: Improving ability for home or yard work: Dissatisfied | 0 | 10 | 1 | 11
  Knee: Improving ability-recreational activities: number analyzed (Participants) | 9 | 58 | 6 | 73
  Knee: Improving ability-recreational activities: Satisfied | 9 | 50 | 5 | 64
  Knee: Improving ability-recreational activities: Dissatisfied | 0 | 8 | 1 | 9
  Hip: Satisfaction with result of surgery: number analyzed (Participants) | 10 | 41 | 6 | 57
  Hip: Satisfaction with result of surgery: Satisfied | 9 | 40 | 6 | 55
  Hip: Satisfaction with result of surgery: Dissatisfied | 1 | 1 | 0 | 2
  Hip: Results of surgery for relieving pain: number analyzed (Participants) | 10 | 41 | 6 | 57
  Hip: Results of surgery for relieving pain: Satisfied | 9 | 41 | 6 | 56
  Hip: Results of surgery for relieving pain: Dissatisfied | 1 | 0 | 0 | 1
  Hip: Improving ability for home or yard work: number analyzed (Participants) | 10 | 41 | 6 | 57
  Hip: Improving ability for home or yard work: Satisfied | 9 | 41 | 6 | 56
  Hip: Improving ability for home or yard work: Dissatisfied | 1 | 0 | 0 | 1
  Hip: Improving ability-recreational activities: number analyzed (Participants) | 10 | 41 | 6 | 57
  Hip: Improving ability-recreational activities: Satisfied | 9 | 40 | 6 | 55
  Hip: Improving ability-recreational activities: Dissatisfied | 1 | 1 | 0 | 2
  Shoulder: Satisfaction with result of surgery: number analyzed (Participants) | 0 | 0 | 1 | 1
  Shoulder: Satisfaction with result of surgery: Satisfied | 0 | 0 | 1 | 1
  Shoulder: Satisfaction with result of surgery: Dissatisfied | 0 | 0 | 0 | 0
  Shoulder: Results of surgery for relieving pain: number analyzed (Participants) | 0 | 0 | 1 | 1
  Shoulder: Results of surgery for relieving pain: Satisfied | 0 | 0 | 1 | 1
  Shoulder: Results of surgery for relieving pain: Dissatisfied | 0 | 0 | 0 | 0
  Shoulder: Improving ability for home or yard work: number analyzed (Participants) | 0 | 0 | 1 | 1
  Shoulder: Improving ability for home or yard work: Satisfied | 0 | 0 | 1 | 1
  Shoulder: Improving ability for home or yard work: Dissatisfied | 0 | 0 | 0 | 0
  Shoulder:Improving ability-recreational activities: number analyzed (Participants) | 0 | 0 | 1 | 1
  Shoulder:Improving ability-recreational activities: Satisfied | 0 | 0 | 1 | 1
  Shoulder:Improving ability-recreational activities: Dissatisfied | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Post-Surgical Complications Upto Week 24
Description: Post-surgical complications are adverse events occurring after TJR surgery that were considered clinically significant as assessed by investigator and attributable to the total joint replacement procedure. Participants may have been counted more than once if they had TJR surgery in more than one joint.
Time Frame: Baseline up to Week 24
Population: Safety analysis set: enrolled participants who had received at least one dose of SC study medication during studies A4091056, A4091057 or A4091058, and who had a qualifying TJR surgery. 'n' = participants evaluable for this OM at specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab Combined | NSAID | All Participants
Number analyzed (Participants) | 20 | 113 | 17 | 150
Participants
  Knee: number analyzed (Participants) | 10 | 66 | 9 | 85
  Knee | 0 | 1 | 0 | 1
  Hip: number analyzed (Participants) | 10 | 48 | 7 | 65
  Hip | 0 | 5 | 0 | 5
  Shoulder: number analyzed (Participants) | 0 | 0 | 1 | 1
  Shoulder | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Additional or Corrective Procedures Related to Total Joint Replacement Upto Week 24
Description: Participants were asked whether they had been told by their orthopedic surgeon that additional or corrective procedures were necessary for their total joint replacement. Participants, who responded as yes have been reported here. Participants may have been counted more than once if they had TJR surgery in more than one joint.
Time Frame: Baseline up to Week 24
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab Combined | NSAID | All Participants
Number analyzed (Participants) | 20 | 113 | 17 | 150
Participants
  Knee: number analyzed (Participants) | 10 | 66 | 9 | 85
  Knee | 0 | 4 | 0 | 4
  Hip: number analyzed (Participants) | 10 | 48 | 7 | 65
  Hip | 0 | 5 | 1 | 6
  Shoulder: number analyzed (Participants) | 0 | 0 | 1 | 1
  Shoulder | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants Who Participated in Physical Rehabilitation Activities Related to Total Joint Replacement Upto Week 24
Description: Participants responded with a yes or no to the following question ''are you participating in physical rehabilitation activities related to your replaced joint''. Participants responded with a yes, have been reported here. Participants may have been counted more than once if they had TJR surgery in more than one joint.
Time Frame: Baseline up to Week 24
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab Combined | NSAID | All Participants
Number analyzed (Participants) | 20 | 113 | 17 | 150
Participants
  Knee: number analyzed (Participants) | 10 | 66 | 9 | 85
  Knee | 10 | 55 | 7 | 72
  Hip: number analyzed (Participants) | 10 | 48 | 7 | 65
  Hip | 9 | 33 | 3 | 45
  Shoulder: number analyzed (Participants) | 0 | 0 | 1 | 1
  Shoulder | 0 | 0 | 1 | 1

6. Primary Outcome: Change From Baseline in Average Pain Score in to be Replaced or Replaced Joints at Week 24
Description: Participants assessed their average pain in to be replaced (pre-surgery) knee/ hip joint or in the replaced joint (post-surgery) in the past 24 hours using an 11-point numerical rating scale (NRS), ranging from 0 (no pain) to 10 (worst possible pain). Higher scores indicated higher pain. Change from baseline was calculated using the difference between post-baseline weekly mean and the baseline mean score. Participants may have been counted more than once if they had TJR surgery in more than one joint.
Time Frame: Baseline, Week 24
Population: Safety analysis set: enrolled participants who had received at least one dose of SC study medication during studies A4091056, A4091057 or A4091058, and who had a qualifying TJR surgery. Here, 'n' = participants evaluable for this OM at specified categories.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: total joint replacements
Arm/Group | Placebo | Tanezumab Combined | NSAID | All Participants
Number analyzed (Participants) | 20 | 113 | 17 | 150
Number analyzed (total joint replacements) | 20 | 113 | 17 | 150
units on a scale
  Baseline: Knee: number analyzed (Participants) | 10 | 71 | 10 | 91
  Baseline: Knee: number analyzed (total joint replacements) | 10 | 71 | 10 | 91
  Baseline: Knee | 6.00 (2.31) | 6.86 (2.14) | 6.80 (2.20) | 6.76 (2.16)
  Baseline: Hip: number analyzed (Participants) | 10 | 48 | 7 | 65
  Baseline: Hip: number analyzed (total joint replacements) | 10 | 48 | 7 | 65
  Baseline: Hip | 6.10 (2.13) | 6.81 (2.27) | 5.86 (3.44) | 6.60 (2.38)
  Change at Week 24: Knee: number analyzed (Participants) | 9 | 63 | 7 | 79
  Change at Week 24: Knee: number analyzed (total joint replacements) | 9 | 63 | 7 | 79
  Change at Week 24: Knee | -4.56 (1.24) | -5.32 (2.63) | -5.43 (2.51) | -5.24 (2.49)
  Change at Week 24: Hip: number analyzed (Participants) | 10 | 42 | 6 | 58
  Change at Week 24: Hip: number analyzed (total joint replacements) | 10 | 42 | 6 | 58
  Change at Week 24: Hip | -5.20 (2.30) | -5.67 (2.37) | -5.00 (4.10) | -5.52 (2.53)

7. Primary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale at Week 24
Description: WOMAC: Self-administered, disease-specific questionnaire, which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis (OA). The WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to OA of to be replaced/replaced index joint (knee or hip) during past 48 hours. It was calculated as the mean of scores from 5 individual questions. Scores for each question and WOMAC Pain subscale score on NRS ranged from 0 (no pain) to 10 (extreme pain), where higher scores indicated higher pain. Change from baseline was calculated using the difference between post-baseline weekly mean and the baseline mean score. Participants may have been counted more than once if they had TJR surgery in more than one joint.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: total joint replacements
Arm/Group | Placebo | Tanezumab Combined | NSAID | All Participants
Number analyzed (Participants) | 20 | 113 | 15 | 148
Number analyzed (total joint replacements) | 20 | 113 | 15 | 148
units on a scale
  Baseline: Knee: number analyzed (Participants) | 10 | 68 | 9 | 87
  Baseline: Knee: number analyzed (total joint replacements) | 10 | 68 | 9 | 87
  Baseline: Knee | 4.66 (3.05) | 5.62 (2.33) | 6.11 (2.31) | 5.56 (2.41)
  Baseline: Hip: number analyzed (Participants) | 10 | 46 | 6 | 62
  Baseline: Hip: number analyzed (total joint replacements) | 10 | 46 | 6 | 62
  Baseline: Hip | 4.80 (2.61) | 5.97 (2.46) | 6.13 (1.98) | 5.80 (2.45)
  Change at Week 24: Knee: number analyzed (Participants) | 9 | 61 | 7 | 77
  Change at Week 24: Knee: number analyzed (total joint replacements) | 9 | 61 | 7 | 77
  Change at Week 24: Knee | -3.13 (1.74) | -4.50 (2.43) | -4.54 (3.15) | -4.34 (2.44)
  Change at Week 24: Hip: number analyzed (Participants) | 10 | 40 | 5 | 55
  Change at Week 24: Hip: number analyzed (total joint replacements) | 10 | 40 | 5 | 55
  Change at Week 24: Hip | -4.34 (2.52) | -4.92 (2.62) | -5.92 (2.40) | -4.91 (2.57)

8. Primary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Subscale at Week 24
Description: WOMAC: self-administered, disease-specific questionnaire, which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with OA. Stiffness was defined as a sensation of decreased ease of movement in the index joint (knee or hip). The WOMAC stiffness subscale is a 2-item questionnaire used to assess the amount of stiffness experienced due to OA in the replaced/to be replaced index joint (knee or hip) during the past 48 hours. It was calculated as the mean of scores from 2 individual questions scored on NRS. Scores for each question and WOMAC stiffness subscale score on NRS ranged from 0 (no stiffness) to 10 (extreme stiffness), where higher scores indicated higher stiffness. Change from baseline was calculated using the difference between post-baseline weekly mean and the baseline mean score. Participants may have been counted more than once if they had TJR surgery in more than one joint.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: total joint replacements
Arm/Group | Placebo | Tanezumab Combined | NSAID | All Participants
Number analyzed (Participants) | 20 | 113 | 15 | 148
Number analyzed (total joint replacements) | 20 | 113 | 15 | 148
units on a scale
  Baseline: Knee: number analyzed (Participants) | 10 | 68 | 9 | 87
  Baseline: Knee: number analyzed (total joint replacements) | 10 | 68 | 9 | 87
  Baseline: Knee | 4.80 (2.78) | 5.75 (2.52) | 6.44 (2.58) | 5.71 (2.55)
  Baseline: Hip: number analyzed (Participants) | 10 | 46 | 6 | 62
  Baseline: Hip: number analyzed (total joint replacements) | 10 | 46 | 6 | 62
  Baseline: Hip | 4.70 (2.75) | 5.96 (2.69) | 5.25 (3.50) | 5.69 (2.77)
  Change at Week 24: Knee: number analyzed (Participants) | 9 | 61 | 7 | 77
  Change at Week 24: Knee: number analyzed (total joint replacements) | 9 | 61 | 7 | 77
  Change at Week 24: Knee | -1.78 (1.52) | -4.13 (2.58) | -3.43 (3.13) | -3.79 (2.62)
  Change at Week 24: Hip: number analyzed (Participants) | 10 | 40 | 5 | 55
  Change at Week 24: Hip: number analyzed (total joint replacements) | 10 | 40 | 5 | 55
  Change at Week 24: Hip | -4.00 (2.66) | -4.48 (2.87) | -3.80 (3.70) | -4.33 (2.86)

9. Primary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale at Week 24
Description: WOMAC: Self-administered, disease-specific questionnaire, which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with OA. Physical function refers to participant's ability to move around and perform usual activities of daily living. The WOMAC physical function subscale is a 17-item questionnaire used to assess the degree of difficulty experienced due to OA in replaced/ to be replaced index joint (knee or hip) during past 48 hours. It was calculated as mean of the scores from 17 individual questions, which may not be a whole (integer) number, scored on a NRS. Scores for each question and WOMAC physical function subscale score on NRS ranged from 0 (no difficulty) to 10 (extreme difficulty), where higher scores indicated extreme difficulty/worse physical function. Participants may have been counted more than once if they had TJR surgery in more than one joint.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: total joint replacements
Arm/Group | Placebo | Tanezumab Combined | NSAID | All Participants
Number analyzed (Participants) | 20 | 113 | 15 | 148
Number analyzed (total joint replacements) | 20 | 113 | 15 | 148
units on a scale
  Baseline: Knee: number analyzed (Participants) | 10 | 68 | 9 | 87
  Baseline: Knee: number analyzed (total joint replacements) | 10 | 68 | 9 | 87
  Baseline: Knee | 4.83 (2.99) | 5.82 (2.11) | 6.63 (1.98) | 5.79 (2.23)
  Baseline: Hip: number analyzed (Participants) | 10 | 46 | 6 | 62
  Baseline: Hip: number analyzed (total joint replacements) | 10 | 46 | 6 | 62
  Baseline: Hip | 5.56 (2.21) | 6.50 (2.22) | 6.86 (1.48) | 6.38 (2.17)
  Change at Week 24: Knee: number analyzed (Participants) | 9 | 61 | 7 | 77
  Change at Week 24: Knee: number analyzed (total joint replacements) | 9 | 61 | 7 | 77
  Change at Week 24: Knee | -2.69 (1.51) | -4.42 (2.19) | -4.59 (2.90) | -4.24 (2.24)
  Change at Week 24: Hip: number analyzed (Participants) | 10 | 40 | 5 | 55
  Change at Week 24: Hip: number analyzed (total joint replacements) | 10 | 40 | 5 | 55
  Change at Week 24: Hip | -4.64 (2.13) | -5.05 (2.44) | -5.95 (1.84) | -5.06 (2.33)

10. Primary Outcome: Change From Baseline in Shoulder Pain and Disability Index (SPADI) Score at Week 24
Description: SPADI: self-administered questionnaire to measure pain and disability associated with shoulder pathology in participants with shoulder pain. It consists of two dimensions pain and function. Pain dimension:5 questions regarding severity of pain, scores ranged from 0=no pain to 10=worst pain imaginable, higher scores indicated extreme pain. Functional activities:8 questions to measure degree of difficulty with various activities of daily living that require upper extremity use, scores ranged from 0=no difficulty to 10=so difficult it requires help, higher scores=extreme difficulty. Pain and disability dimension score was calculated as the sum of non-missing scores divided by the maximum possible score (50 [for pain] and 80 [for disability]) multiplied by 100. A total score was calculated as the mean of two dimensions, ranged from 0=best to 100=worst, higher scores indicated worsening of condition.
Time Frame: Baseline, Week 24
Population: Enrolled participants who received at least one dose of SC study medication during studies A4091056, A4091057 or A4091058, and who had qualifying shoulder replacement. "N"=those participants who had data available for this OM, hence data for Placebo and Tanezumab reporting groups were not collected as no participants were evaluable for this OM.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: total joint replacements
Arm/Group | Placebo | Tanezumab Combined | NSAID | All Participants
Number analyzed (Participants) | 0 | 0 | 1 | 1
Number analyzed (total joint replacements) | 0 | 0 | 1 | 1
units on a scale
  Baseline |  |  | 89.88 | 89.88
  Change at Week 24 |  |  | -89.88 | -89.88

11. Primary Outcome: Number of Participants Who Used Concomitant Analgesic Medications
Time Frame: Baseline up to Week 24
Population: Safety analysis set: all enrolled participants of this study who had received at least one dose of SC study medication during studies A4091056, A4091057 or A4091058, and who had a qualifying TJR surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab Combined | NSAID | All Participants
Number analyzed (Participants) | 20 | 113 | 17 | 150
Participants | 18 | 100 | 15 | 133

ADVERSE EVENTS:
Time Frame: Baseline up to Week 24
Description: Same event may appear as both an adverse event (AE) and serious AE. What is presented are distinct events. An event may be categorized as serious in one and as non-serious in another or one participant may have experienced both serious and non-serious event. Safety set analyzed. AEs for tanezumab were collected and reported dose wise and combined.
Groups:
- Tanezumab 2.5 mg: Participants who received tanezumab 2.5 mg SC injection in studies A4091056, A4091057 or A4091058 and who had undergone a TJR surgery, were followed up for a maximum duration of 24 weeks in this study. Baseline for this study was the last visit in study A4091056, A4091057 or A4091058 or when the site notified of a planned TJR surgery.
- Tanezumab 2.5/5 mg: Participants who received tanezumab 2.5/5 mg SC injection in study A4091056 and who had undergone a TJR surgery, were followed up for a maximum duration of 24 weeks in this study. Baseline for this study was the last visit in study A4091056, A4091057 or A4091058 or when the site notified of a planned TJR surgery.
- Tanezumab 5 mg: Participants who received tanezumab 5 mg SC injection in studies A4091057 or A4091058 and who had undergone a TJR surgery, were followed up for a maximum duration of 24 weeks in this study. Baseline for this study was the last visit in study A4091056, A4091057 or A4091058 or when the site notified of a planned TJR surgery.
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg | Tanezumab 5 mg | Tanezumab Combined | NSAID | All Participants
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/52 | 0/8 | 0/53 | 0/113 | 0/17 | 0/150
Serious Adverse Events (participants affected / at risk) | 0/20 | 5/52 | 3/8 | 7/53 | 15/113 | 2/17 | 17/150
Other Adverse Events (participants affected / at risk) | 0/20 | 9/52 | 3/8 | 9/53 | 21/113 | 4/17 | 25/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=20) | Tanezumab 2.5 mg (N=52) | Tanezumab 2.5/5 mg (N=8) | Tanezumab 5 mg (N=53) | Tanezumab Combined (N=113) | NSAID (N=17) | All Participants (N=150)
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 1
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 3 | 2 | 5
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 0 | 1
Parkinson's disease (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Device dislocation (Product Issues) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=20) | Tanezumab 2.5 mg (N=52) | Tanezumab 2.5/5 mg (N=8) | Tanezumab 5 mg (N=53) | Tanezumab Combined (N=113) | NSAID (N=17) | All Participants (N=150)
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 6 | 9 | 0 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 3 | 0 | 3
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0 | 3 | 0 | 3
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 2 | 0 | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 2
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 2 | 0 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-01-06): https://cdn.clinicaltrials.gov/large-docs/86/NCT02674386/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-02): https://cdn.clinicaltrials.gov/large-docs/86/NCT02674386/SAP_001.pdf